CLINICAL TRIAL: NCT05251844
Title: Effectiveness of Email Alerting on Reducing Hospital Employees' Unauthorized Access to Protected Health Information: A Nonrandomized Controlled Trial
Brief Title: The Effectiveness of Email Alerting on Reducing Employees' Unauthorized Access to Protected Health Information
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Protenus, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: email_alert_effectiveness
Record Dates: First submitted 2022-02-01; First posted 2022-02-23 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Unauthorized Data Access

STUDY DESIGN:
Intervention Model Description: one group received email notice while the group didn't
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: all violators' identities are masked to Protenus.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Email warning (Experimental): some individuals that accessed patients' data without authorization were randomly selected to receive an email warning. A sample email:
  Dear Colleague,
  The {Organization} proactive electronic record monitoring system has flagged you as having accessed the electronic patient record of {Patient_Name} on {Case_Event_Date}. A clear work-related purpose has not been identified for this access, and there are no approvals in place by the {Organization} Privacy Office to allow access to this record for personal purposes in accordance with A065. {Organization} takes the privacy of patient information very seriously. The {Organization} Privacy Office is now investigating this access as a potential privacy breach.
  This potential noncompliance needs to be resolved immediately. To help determine whether a privacy breach has occurred, please respond to this email with answers to the following questions no later than 5 days from the date of this email...omitted due to length
  Interventions: Other: receiving an email
- No eamil warning (No Intervention): individuals that were flagged as accessing patients' data without authorization on the same day as the experimental group were used as the control group

INTERVENTIONS:
Other: receiving an email — The email informed that the employee has had been identified as having accessed a patient's electronic medical record without a known work-related purpose and that unauthorized access is a privacy violation.
  Arms: Email warning

SUMMARY:
To assess the effectiveness of email warnings on reducing repeated unauthorized access to Protected Health Information (PHI), a randomized trial was conducted in a large academic medical center to understand the effectiveness of email warning on reducing repeated unauthorized access to PHI.

DETAILED DESCRIPTION:
From January 1, 2018, to July 31, 2018, a large academic medical center's PHI access monitoring system flagged all unauthorized accesses to patient electronic medical records from 444 employees (all professional medical staff), who were not part of the patient's intervention team and did not have access permission. 219 employees (49%) were randomly selected to receive an email warning on the night of their access, while the remaining employees (225, 51%) served as controls. The email informed that the employee has had been identified as having accessed a patient's electronic medical record without a known work-related purpose and that unauthorized access is a privacy violation. A sample email was attached at the end of the protocol.

The system tracked all these individuals' violations within the sample period. Later on, all cases with the violators' ID and patients' ID fully de-identified (see the following excerpt as examples) were shared with researchers at John Hopkins and Michigan State for data analyses. Because researchers do not have the ability to link the data with an identifier, the study was exempted from Michigan State University's IRB review.

Violator ID Patient ID Date Intervention 01B1NSYX3CEXZ86UZXU7R9JQ4VEK R7Z8RTZQL4B9IAC13F6EXQJVWAI7 1/2/2018 No Email

01B1NSYX3CEXZ86UZXU7R9JQ4VEK R7Z8RTZQL4B9IAC13F6EXQJVWAI7 1/3/2018 No Email

ELIGIBILITY:
Inclusion Criteria:

* violators of patients' privacy rights

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 444 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
the number of subsequent unauthorizated access violations | 12 weeks starting from the first time a violation was flagged
  The investigators monitored and collected all the subsequent unauthorized access violations for both the experiment and the control group

CONTACTS AND LOCATIONS:
Overall Officials: Nick Culbertson, BS, Study Chair — Protenus, Inc.
Locations (1):
- Protenus, Inc., Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
The data were collected from a large academic medical center that wanted to remain anonymous